CLINICAL TRIAL: NCT01843127
Title: A Phase 1, Randomized, Single-blind, Placebo-controlled, Multiple-dose, Two-sequence, Cross-over Study to Evaluate the Effect of Ranolazine on Glucagon Secretion in Subjects With Type 2 Diabetes Mellitus, Followed by An Open-label, Single Dose, Exenatide Active-control Period
Brief Title: A Study to Evaluate the Effect of Ranolazine on Postprandial Glucagon in Subjects With Type 2 Diabetes.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GS-US-259-0165
Record Dates: First submitted 2013-04-17; First posted 2013-04-30 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ranolazine; Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo, Ranolazine, Exenatide (Active Comparator)
  Interventions: Drug: Ranolazine; Drug: Placebo; Drug: Exenatide
- Ranolazine, Placebo, Exenatide (Active Comparator)
  Interventions: Drug: Ranolazine; Drug: Placebo; Drug: Exenatide

INTERVENTIONS:
Drug: Ranolazine
Drug: Placebo
Drug: Exenatide

SUMMARY:
To explore the mechanism of action of ranolazine as a potential treatment for type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 65 years old, inclusive
* Documented history of T2DM for ≥5 years
* Body mass index (BMI) 20.0 to 40.0 kg/m2, inclusive, at Screening
* Stable treatment (≥ 12 weeks) with metformin alone, a sulfonylurea alone, a meglitinide alone, or a combination of metformin with either a sulfonylurea or a meglitinide
* HbA1c ≥ 7.0% and ≤ 10.5%, inclusive, at Screening
* Fasting glucose within specific ranges, at Screening and after 14 +/-2 days of wash-out from prior oral anti-diabetic agents
* Fasting serum C-peptide ≥0.8 ng/mL, at Screening
* Estimated glomerular filtration rate (eGFR)≥60 mL/min/1.73 m2
* Ability and willingness to comply with all study procedures during the course of the study, including washout from oral anti-diabetic (OAD) agents approximately 2 weeks prior to Day -2 admission
* Females of childbearing potential must have a negative pregnancy test at Screening and on Day -2 admission and must agree to use highly effective contraception methods from Screening throughout study participation and for 14 days following the last dose of study drug.

Exclusion Criteria:

* History of type 1 diabetes mellitus or secondary forms of diabetes
* History of acute diabetes complications
* Recent or significant heart conditions
* Uncontrolled hypertension
* QTc interval > 500 msec by ECG at Screening or on Day -2 admission, a personal or family history of QTc prolongation, congenital long QT syndrome, or use of drugs that prolong the QTc interval, such as Class Ia or Class III antiarrhythmic agents, erythromycin, and certain antipsychotics (eg, ziprasidone)
* History of severe GI disease (e.g., gastroparesis)
* History of pancreatitis (acute or chronic)
* Current consumption of > 14 alcoholic drinks per week, or more than 4 alcoholic drinks on any one day
* Current regular use of tobacco- or nicotine-containing products in excess of 10 cigarettes per day or equivalent
* History of substance abuse within 12 months prior to Screening
* Significant hepatic disease, including, but not limited to, chronic active hepatitis and liver cirrhosis (Child-Pugh Class A, B, or C)
* History of malignancy within 5 years prior to Screening
* Significant thyroid disease
* Treatment with selected medications, as indicated in the protocol
* Prior treatment with open-label ranolazine or known hypersensitivity or intolerance to ranolazine or its excipients
* Known hypersensitivity or intolerance to GLP-1 mimetics
* Known hypersensitivity or intolerance to acetaminophen
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 X upper limit of normal (ULN)
* Total Bilirubin (TB) > 2 mg/dL
* Hemoglobin < 12 g/dL (for males) or < 11 g/dL (for females)
* Positive for hepatitis B surface antigen
* Positive for anti-hepatitis C virus antibody
* Positive for human immunodeficiency virus-1 (HIV-1) antibody
* Positive urine drug screen
* Positive alcohol test
* Donation of blood or blood products to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 500 mL of blood during the 6 weeks prior to Screening
* Females who are pregnant or breastfeeding
* Other condition(s) that, in the opinion of the investigator, would compromise the safety of the subject, would prevent compliance with the study protocol, or would compromise the quality of the clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) of plasma glucagon during the standard meal test (SMT) | Days 5, 10, and 14

SECONDARY OUTCOMES:
Plasma glucose, serum insulin, and serum C-peptide AUCs during the SMT | Days 5, 10, and 14
Collapse under Acetaminophen PK | Days 5 and 10
Area under the plasma acetaminophen concentration-time curve from time 0 to 240 min (AUC0-240 min) | Days 5 and 10
Collapse all under ranolazine pharmacokinetics (PK) | Days 5 and 10
Trough plasma ranolazine concentrations (Ctrough) | Days 5 and 10
Average plasma ranolazine concentration during a dosing interval at steady state (Css,ave) | Days 5 and 10
Area under the plasma ranolazine concentration-time curve over dosing interval (AUCtau) | Days 5 and 10
Apparent elimination half-life (t1/2) of ranolazine | Days 5 and 10
Adverse events, physical examinations, clinical laboratory determinations, electrocardiograms (ECG), and vital sign assessments. | From Screening to 7 days after the final dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - SeaView Research, Inc, Miami, Florida
  - Translational Research Institute-Florida Hospital, Orlando, Florida